CLINICAL TRIAL: NCT05554913
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Phase 3 Study Evaluating the Efficacy and Safety of Recombinant Human Thrombopoietin Mimetic Peptide-Fc Fusion Protein for Injection (QL0911) in the Prevention of Chemotherapy- Induced Thrombocytopenia
Brief Title: Evaluating the Efficacy and Safety of QL0911 in the Prevention of Chemotherapy- Induced Thrombocytopenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QL0911-CIT-301(Part B)
Record Dates: First submitted 2022-09-18; First posted 2022-09-26 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2022-09

CONDITIONS: Chemotherapy-induced Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL0911 (Experimental): The study in a 2:1 randomization ratio(40 subjects to QL0911). Qilu investigational product (QL0911 or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Interventions: Drug: QL0911
- Placebo (Placebo Comparator): The study in a 2:1 randomization ratio(20 subjects to Placebo ). Qilu investigational product (QL0911 or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QL0911 — This study is designed to study QL0911 for the treatment of chemotherapy-induced thrombocytopenia (CIT) in patients receiving chemotherapy for cancer
  Arms: QL0911
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of QL0911 to prevention chemotherapy-induced thrombocytopenia. Thrombocytopenia is a low number of platelets in the blood. Sometimes, thrombocytopenia occurs as a side effect of chemotherapy treatments.

DETAILED DESCRIPTION:
For the phase III study, a double-blind randomized, placebo controlled, parallel-group design will be conducted to evaluate the efficacy and safety of QL0911 . Each subject will be randomly assigned to either Arm A (QL0911) or Arm B (placebo) in 2:1 ratio.The primary objective is to compare the effective rates of the two treatment arms. The study will consist of a screening period of up to 4 weeks, a treatment period of 2 planned cycles of chemotherapy, a follow-up visit of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old;
* Histopathological or cytological examination confirmed solid tumor or lymphoma (including NSCLC, breast cancer, bladder cancer, pancreatic cancer, etc.), chemotherapy cycle of 21 days, and using of one or more of the following chemotherapy drugs: gemcitabine; Platinum, including carboplatin, nedaplatin, cisplatin, lobaplatin, etc.; Anthracyclines, including doxorubicin, daunorubicin, epirubicin, etc.; Taxa, including paclitaxel, docetaxel, etc.
* The current chemotherapy regimen should be consistent with that of the previous chemotherapy cycle, including the chemotherapy drugs and the dosages, without adding or subtracting drugs or dosages;
* At least two platelet counts with an interval of more than 24 hours in the chemotherapy cycle before enrollment was grade 2 or higher thrombocytopenia;
* The platelet count was between 75×10^9/L-150×10^9/L (including both ends) 1 day before chemotherapy or the day of Randomization;
* At the time of screening, the expected survival time is ≥12 weeks, and the current chemotherapy regimen can be accepted for at least 2 cycles;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2;
* Fully understand and comply with the requirements of this study, and voluntarily sign the informed consent form.

Exclusion Criteria:

* Suffering from other hematopoietic system diseases besides lymphoma, including leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma and myelodysplastic syndromes, etc.
* Have experienced thrombocytopenia caused by non-tumor chemotherapeutics within 6 months before screening,Including, but not limited to, EDTA-dependent pseudothrombocytopenia, hypersplenism, infection, and bleeding, etc.
* Brain tumors, brain metastases,bone marrow invasion or bone marrow metastasis;
* Receiving radiotherapy or have received abdominal pelvic or sternum radiotherapy within 3 months;
* Any arterial or venous thrombosis occurred within 6 months before screening;
* Severe cardiovascular disease (e.g., NYHA Heart Function Score Class III-IV), arrhythmias such as atrial fibrillation that increase the risk of thrombosis, coronary stenting, angioplasty, and coronary artery bypass grafting within the previous 6 months were screened;
* Clinical manifestations of severe bleeding (such as gastrointestinal bleeding, etc.) within 4 weeks before the first administration of the experimental drug;
* Received platelet transfusion within 5 days before randomization/enrollment;
* Received thrombopoietin receptor agonist treatment within 4 weeks, human recombinant thrombopoietin (rhTPO) or rhIL-11 within 4 weeks,other Chinese medicines with the effect of raising blood plate within 1 week before the administration of the experimental drug;
* Used heparin, warfarin, aspirin and other anticoagulant drugs within 7 days before the first dose except for the purpose of sealing the tube;
* Received bone marrow transplantation or stem cell infusion within 1 year before screening;
* Patients with hepatitis C antibody positive and detection of HCV-RNA exceeding the upper limit, patients with hepatitis B surface antigen positive and detection of HBV-DNA exceeding the upper limit, patients with severe cirrhosis, HIV antibody positive and syphilis antibody positive;
* The absolute value of neutrophils in the screening period<1.5×10^9/L, hemoglobin <90g/L;
* Total bilirubin greater than 3X ULN; alanine aminotransferase [ALT] and aspartate aminotransferase [AST] greater than 3X ULN for subjects without liver metastases or greater than or equal to 5X ULN for subjects with liver metastases during screening;
* Serum creatinine concentration ≥1.5ULN or eGFR≤45ml/min (cockcroft-gault);
* Severe drug allergic reactions;
* Used any investigational drug within 3 months before the administration of the experimental drug;
* Planning pregnancy, pregnancy, or suckling period;
* The investigator judged that the patients are not suitable for participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who had an efficacy response during the double-blind period | 42 days

SECONDARY OUTCOMES:
Lowest and highest platelet count | 42 days
Bleeding score(Revised WHO grading system) | 42 days
Proportion of patients with platelet count < 50×10^9/L per cycle | 42 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China